CLINICAL TRIAL: NCT05658328
Title: A Neighborhood-based Physical and Social Activity Intervention for Older Black Caregivers and People Living With Dementia: SHARP-CG
Brief Title: Neighborhood-based Physical and Social Activity for Older Black Caregivers and People Living With Dementia
Acronym: SHARP-CG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Raina Croff, Assistant Professor of Neurology, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 5P30AG024978-19 (NIH); P30AG024978-19 (NIH)
Record Dates: First submitted 2022-11-11; First posted 2022-12-20 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Caregiver Burden; Depression; Cognitive Impairment
Keywords: physical activity; reminiscence; social engagement; dementia caregiver; neighborhood-based; walking; technology-enabled; sleep; geriatric depression; caregiver burden; African American
MeSH Terms: conditions — Caregiver Burden; Depression; Cognitive Dysfunction; Motor Activity

STUDY DESIGN:
Intervention Model Description: Triads are randomized into either the intervention group or the waitlist control group. The intervention group walks for 16 weeks. The waitlist control group completes baseline measures for 16 weeks then continues measures while walking 16 weeks. Wearable technology and weekly surveys are optional for PLWD.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Caregivers (MCI or healthy) randomized into this group walk 3x/week for 16 weeks with their care-partner (person living with early-stage dementia - PLWD) and their caregiver support person (MCI or healthy). Caregivers (and optionally for PLWD), wears an actigraphy watch, uses an under-the-mattress sleep sensor, and on a weekly basis completes weight and a health update survey. Mid- and end-study focus groups evaluate program effectiveness and needed adaptations.
  Interventions: Behavioral: SHARP - Physical and social activity
- Waitlist Control (Active Comparator): Caregivers (MCI or healthy) randomized into this group first complete baseline measures for 16 weeks, consisting of wearing an actigraphy watch, using an under-the-mattress sleep sensor, and, on a weekly basis, completing weight and a health update survey. These baseline measures are optional for PLWD. After 16 weeks of baseline data collection, the primary caregiver continues these measures while walking 3x/week for 16 weeks with their triad. The PLWD optionally completes measures and optionally wears the watch and sleep sensor. Mid- and end-study focus groups during the walking phase evaluate program effectiveness and needed adaptations.
  Interventions: Behavioral: SHARP - Physical and social activity

INTERVENTIONS:
Behavioral: SHARP - Physical and social activity — Technology-enabled neighborhood walking 3x/week for 16 weeks with conversational reminiscence

SUMMARY:
The Sharing History through Active Reminiscence and Photo-imagery (SHARP) Program engages triads (primary caregiver, person living with dementia, caregiver support person) in walking and social reminiscence, using a group tablet to access routes and historical neighborhood images serving as conversational prompts. Focus is on adapting the SHARP model to older Black dementia caregivers and on caregiver physical and mental health. Study technology measures sleep and daily step count. Weekly online surveys assess health status. Pre-post assessments measure cognitive function and mental health. Focus groups assess adaptation needs, feasibility and acceptance, and cultural significance.

DETAILED DESCRIPTION:
The Sharing History through Active Reminiscence and Photo-imagery (SHARP) Program is a recently developed culturally celebratory, multimodal approach to physical, social, and reminiscence activity. The SHARP walking application, accessed on a group tablet, is preloaded with 72 themed, 1-mile neighborhood routes with GPS-linked "Memory Markers," historical neighborhood images and questions, to prompt conversational reminiscence about Black life, history, and culture. In this Stage I study, walking triads consist of a healthy or mildly cognitively impaired (MCI) primary dementia caregiver (aged 55+), the care partner - a person living with early-stage dementia (PLWD) or MCI (aged 55+), and a healthy or MCI caregiver support person (aged 18+). Triads walk 3x/week over 16 weeks in the gentrifying, historically Black neighborhoods of Portland, Oregon. The primary caregiver wears an actigraphy watch, uses an under-the-mattress sleep sensor, and on a weekly basis, measures weight on a study-provided digital scale and completes a health update survey. Watch, sleep sensor, and weekly measures are optional for the PLWD. We aim to (1) adapt SHARP implementation, technology, and protocol for caregivers of PLWD, and (2) test preliminary efficacy of this intervention on dementia caregivers' physical and mental health.

ELIGIBILITY:
Inclusion Criteria:

1. Self-identified African American (caregiver and PWD)
2. Caregivers and PWD Age > 55 years old; caregiver support person aged >18 years old
3. Caregiver and PWD reside or resided for >10 years in Portland's historically Black neighborhoods (to be familiar with Memory Markers about this area)
4. Able to ambulate independently for at least 45 minutes without the use of mobility aids
5. Meeting Cognition Criteria

   a. Participants with MCI or early-stage/mild dementia will meet criteria consistent with those defined by Jak et al. and with the criteria outlined by the NIA-Alzheimer's Association workgroup
6. Cognitive function allows independent (or minimally assisted) travel to and from walk locations
7. Caregivers must have in-home reliable broadband internet (for weekly online surveys).
8. Ability to read, speak, and understand English - all participants
9. In general good health for their age (e.g., stable cardiovascular disease, stable diabetes mellitus, no significant nervous system disease).
10. Subject must have adequate vision, hearing and language abilities to complete assessments.

Exclusion Criteria:

1. Self-reported or clinically diagnosed late-stage dementia
2. Significant disease of the central nervous system
3. Severely depressed (CES-D score > 16), significantly symptomatic psychiatric disorder
4. Advanced cardiovascular disease that would make walking difficult, including history of congestive heart failure
5. Unstable insulin-dependent diabetes mellitus, received diagnosis Type 1 Diabetes, started insulin within past 3 months, hospitalized for hypoglycemia within past 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-10-20 (Actual); Study Completion 2024-10-20 (Actual)

PRIMARY OUTCOMES:
Effect on sleep health | 16 weeks
  Primary caregivers (and optionally PLWD) continuously wear an actigraphy watch for the study duration. The watch (Withings) measures heart rate variability, step-activity levels, sleep times, and sleep disturbances. Step counts (watch), total sleep time and quality (bed-mat sleep sensor), and HRV (watch and sleep sensor) will be analyzed using generalized mixed effects models with outcome being each incidence of occurrence (e.g., blue mood) or continuous outcomes (e.g., daily duration of sleep) and a time*group interaction term.
Effect on sleep health | 16 weeks
  Primary caregivers (and optionally PLWD) use an under-the-mattress sleep sensor that measures sleep time and quality, HRV, and movement activity. Step counts (watch), total sleep time and quality (bed-mat sleep sensor), and HRV (watch and sleep sensor) will be analyzed using generalized mixed effects models with outcome being each incidence of occurrence (e.g., blue mood) or continuous outcomes (e.g., daily duration of sleep) and a time*group interaction term.
Change in blood pressure | 16 weeks
  Pre-post difference in blood pressure are compared between primary caregivers in the experimental (SHARP intervention) and control groups (i.e., control (usual behavior) group waits 4 months then walks 4 months). Linear regression models with the primary and secondary outcome (BP and ZBI-12 (1°), at month 4 will be regressed on the baseline score of each outcome, the treatment group (experimental vs. control groups), controlling for caregiver age. The coefficient of the treatment group variable indicates the efficacy of the experiment.

SECONDARY OUTCOMES:
Effect on mental health | 16 weeks
  The Short Form Zarit Burden Interview (ZBI-12) is administered pre-post intervention. Pre-post difference in scores are compared between primary caregivers in the experimental (SHARP intervention) and control groups (i.e., control (usual behavior) group waits 4 months then walks 4 months). Linear regression models with the primary and secondary outcome (BP and ZBI-12 (1°), at month 4 will be regressed on the baseline score of each outcome, the treatment group (experimental vs. control groups), controlling for caregiver age. The coefficient of the treatment group variable indicates the efficacy of the experiment.

OTHER OUTCOMES:
Design effectiveness | 16 weeks
  Focus groups evaluate program design effectiveness for older Black dementia caregivers, including acceptance, needed adaptations, and cultural significance

CONTACTS AND LOCATIONS:
Overall Officials: Raina L Croff, PhD, Principal Investigator — OregonOHSU
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Croff RL, Witter Iv P, Walker ML, Francois E, Quinn C, Riley TC, Sharma NF, Kaye JA. Things Are Changing so Fast: Integrative Technology for Preserving Cognitive Health and Community History. Gerontologist. 2019 Jan 9;59(1):147-157. doi: 10.1093/geront/gny069. PMID 29961887
- [Background] Paula Carder, Raina Croff, Aliza Tuttle & Juell Towns (2022) Walking and Talking: Recommendations for Doing Mobile Interviews with Older Adults, Journal of Aging and Environment, DOI: 10.1080/26892618.2022.2030844
- See also: SHARP study website — http://www.sharpwalkingstudy.org